CLINICAL TRIAL: NCT01403012
Title: Differential Analysis of Metabolomic Profiles in Patients With Chronic Plaque Psoriasis Undergoing Systemic Treatment
Brief Title: BOSTRIP: Biomarkers of Systemic Treatment Response in Psoriasis
Acronym: Bostrip
Status: Terminated | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: BOS-1168-WEI-0080-I
Record Dates: First submitted 2011-07-08; First posted 2011-07-27 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis
Keywords: To identify clinical and metabolomic markers that underlie variability in response to systemic therapy in psoriasis; To identify metabolomic signatures associated with psoriasis; To identify possible treatment-specific metabolomic signatures
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Psoriasis patients
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Withdrawal of venous blood samples — Withdrawal of venous blood samples (approx. 20 ml) and 2 skin biopsies (5 mm)
  Laboratory measurements:
  Fasting serum concentrations of 200 metabolites covering a biologically relevant panel of amino acids, sugars, acylcarnitines and phospholipids Genome-wide expression profiles generated from RNA derived from peripheral leukocytes

SUMMARY:
Metabolomics of systemic psoriasis treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 80 years, body weight ≤ 180 kg
* Dermatological diagnosis of psoriasis
* Initiated therapy with TNFα-inhibitor agents (etanercept, adalimumab and infliximab)or fumaric acid ester (FAE) within the scope of routine patient care by treating physician
* Signed informed consent from patient

Exclusion Criteria:

* Patients with evidence of any skin condition that would interfere with the evaluation of psoriasis
* Use of systemic anti-psoriatic drugs such as steroids, retinoids, methotrexate, cyclosporine within 30 days of Visit 1 or used FAE or other any biologic agent such as etanercept, infliximab and adalimumab within 12 weeks prior to Visit 1
* Patients who are considered potentially unreliable or where it is envisaged the patient may not consistently attend scheduled study visits
* Patients who are unable to complete a patient diary or complete questionnaires on paper
* Patients with any other condition or prior/current treatment, which in the opinion of the investigator renders the patient ineligible for the study schedule
* Pregnancy or breast feeding women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant unless they use effective contraception during the study. Effective contraception is defined as either: use of established oral, injected or implanted hormonal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11-19 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
Analysis of metabolic profiles associated with treatment response | week 0 and week 12
  The primary aim of this study is to analyze metabolic profiles as well as expression data in patients with chronic plaque psoriasis undergoing systemic treatment with TNF_-inhibitor agents (etanercept, adalimumab, infliximab) and fumaric acid ester (FAE) in order to identify clinical and metabolomic markers that underlie variability in response to therapy.

SECONDARY OUTCOMES:
Identification of metabolomic signatures associated with psoriasis | week 0 and week 12
  The secondary aim is to identify metabolomic signatures associated with psoriasis and to identify possible treatment-specific metabolomic signatures.
  It is anticipated, to get insights into mechanisms of anti-TNF drug action and response as well as first indications for metabotypes that are associated with psoriasis. In addition, genetic variants correlated to these metabotypes might be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, Dr. med., Principal Investigator — Dermatology, University Kiel
Locations (1):
- Department of Dermatology and Allergy, Uniklinik Kiel, Kiel, Schleswig-Holstein, Germany